CLINICAL TRIAL: NCT05022732
Title: Double-blind, Randomized, Placebo-controlled Clinical Study to Evaluate the Effect on Weight of a Medical Device Based on Polyglucosamine L112® in a Group of Overweight and Obese Subjects
Brief Title: Polyglucosamine L112 in Overweight and Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200037586
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: Obesity; Polyglucosamine; Body composition; Inflammation
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control formula (Placebo Comparator): Excipients and gum arabic in tablet
  Interventions: Combination Product: Placebo
- Experimental formula (Active Comparator): Polyglucosamine L112 (750 mg of chitosan for tablet formulated with ascorbic acid and tartaric acids in the relative proportions of 91-6-3% with the addition of formulating excipients)
  Interventions: Dietary Supplement: Polyglucosamine L112

INTERVENTIONS:
Dietary Supplement: Polyglucosamine L112 — 750 mg of chitosan for tablet formulated with ascorbic acid and tartaric acids in the relative proportions of 91-6-3% with the addition of formulating excipients
  Arms: Experimental formula
Combination Product: Placebo — excipients and gum arabic
  Arms: Control formula

SUMMARY:
This research proposes as its main purpose to evaluate the effectiveness of the intake of Polyglucosamine at a dose of 3 g / day on weight loss in a group of subjects suffering from overweight and mild obesity (BMI between 25 and 32 kg / m2). and with weight> 75 kg

ELIGIBILITY:
Inclusion Criteria:

* weight > 75 Kg
* absence of previous diet therapy attempts
* no fluctuation of at least 3 kg in the previous 3 months
* Beck Depression Inventory score < 20 pt
* Binge Eating Scale score < 27 pt

Exclusion Criteria:

* allergy to shellfish
* pregnancy or breast feeding
* presence of cardiopathies, nephropathies, liver diseases, bronchopneumopathies, haemopathies, dermopathies, chronic-degenerative diseases of the Central Nervous System
* presence of active peptic ulcer, ulcerative colitis, Crohn's disease, celiac disease, inflammatory bowel disease
* symptomatic cholelithiasis
* previous or current neoplasms
* epilepsy
* obesity secondary to endocrinopathies or genetic syndromes
* significant motor disability or mental retardation
* major depressive disorder, bulimia, panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, bipolar disorder (I or II), schizophrenia
* previous history or current diagnosis of drug abuse or alcoholism
* changing in smoking habits or quitting smoking in the last 6 months
* current use or in the last 3 months of psychoactive drugs or current use or in the last 12 months of drugs affecting body weight or appetite

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Changes on anthropometric measures | Changes from baseline anthropometric measures at 90 days
  Body weight (Kg)

SECONDARY OUTCOMES:
Changes on lipid profile | Changes from baseline lipid profile at 90 days
  Total Cholesterol (mg/dl), High Density Lipoprotein Cholesterol (mg/dl), Low Density Lipoprotein Cholesterol (mg/dl), Triglycerides (mg/dl)
Changes on insulin resistance | Changes from baseline insulin resistance at 90 days
  Homeostasis Model Assessment (pt) for evaluate insulin resistance il > 2,4
Changes on Carbohydrate profile | Changes from baseline Carbohydrate profile at 90 days
  Glycemia (mg/dl)
Changes on Carbohydrate profile | Changes from baseline Carbohydrate profile at 90 days
  Insulin (mcU/ml)
Changes on safety | Changes from baseline safety at 90 days
  Aspartate aminotransferase (IU/l), alanine aminotransferase (IU/l)
Changes on safety | Changes from baseline safety at 90 days
  Gamma glutamyl transferase (U/I)
Changes on safety | Changes from baseline safety at 90 days
  Creatinine (mg/dl)
Changes on anthropometric measures | Changes from baseline anthropometric measures at 90 days
  Waist circumference (cm)
Changes on anthropometric measures | Changes from baseline anthropometric measures at 90 days
  Body Mass Index (Kg/m2)
Changes on body composition | Changes from baseline body composition at 90 days
  Free Fat Mass (g), Fat Mass (g), Visceral Adipose Tissue (g)
Changes on oxidative stress | Changes from baseline oxidative stress at 90 days
  Reactive Oxygen Species (CARR U)
Changes on oxidative stress | Changes from baseline oxidative stress at 90 days
  Total Antioxidant Capacity (ORAC U)

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, Principal Investigator — Fondazione Casemiro Mondino
Locations (1):
- Azienda di Servizi alla Persona, Pavia, Italy